CLINICAL TRIAL: NCT05298787
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, SAD/MAD Adaptive-Design Study to Assess the Safety, Tolerability, PK, and PD of RLS-0071 in Healthy Adult Subjects in Support of a COVID-19 Development Program
Brief Title: A Phase 1 SAD/MAD Study of RLS-0071 in Healthy Volunteers in Support of a COVID-19 Development Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReAlta Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLS-0071-101
Record Dates: First submitted 2022-03-15; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — RLS-0071

STUDY DESIGN:
Intervention Model Description: Each cohort will include 8 subjects randomized to receive either RLS-0071 (6 subjects) or placebo (2 subjects). Up to 7 cohorts (4 single-ascending dose [SAD] and 3 multiple-ascending dose [MAD]) enrolling up to 56 subjects are planned for the study. Subjects enrolled in a SAD cohort will receive a single infusion of RLS-0071. Subjects enrolled in a MAD cohort will receive a RLS-0071 infusion every (q) 8 hours for a total of 9 doses, with the ninth infusion occurring in the morning on Day 4. Dose escalation will depend on the Safety Review Committee (SRC) review of available blinded safety and PK data through the observation period of the previous cohort (ie, 48 hours after the last dose of study intervention).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- SAD - 2mg/kg or placebo IV infusion (Experimental): Single IV infusion
  Interventions: Drug: RLS-0071; Drug: Saline Placebo
- SAD - 10mg/kg or placebo IV infusion (Experimental): Single IV infusion
  Interventions: Drug: RLS-0071; Drug: Saline Placebo
- SAD - 40mg/kg or placebo IV infusion (Experimental): Single IV infusion
  Interventions: Drug: RLS-0071; Drug: Saline Placebo
- MAD - 2mg/kg or placebo IV infusion (Experimental): IV infusion given every 8 hours over 3 days for a total of 9 doses
  Interventions: Drug: RLS-0071; Drug: Saline Placebo
- MAD - 10mg/kg or placebo IV infusion (Experimental): IV infusion given every 8 hours over 3 days for a total of 9 doses
  Interventions: Drug: RLS-0071; Drug: Saline Placebo
- SAD - 120mg/kg or placebo IV infusion (Experimental): Single IV infusion
  Interventions: Drug: RLS-0071; Drug: Saline Placebo
- MAD - 40mg/kg or placebo IV infusion (Experimental): IV infusion given every 8 hours over 3 days for a total of 9 doses
  Interventions: Drug: RLS-0071; Drug: Saline Placebo

INTERVENTIONS:
Drug: RLS-0071 — RLS-0071 is administered as an IV infusion
Drug: Saline Placebo — Placebo is administered as an IV infusion

SUMMARY:
This is a Phase 1, single-center, randomized, double-blind, placebo-controlled, adaptive-design study to assess the safety, tolerability, PK, and PD of single- and multiple-ascending doses of RLS-0071 in healthy adult subjects.

DETAILED DESCRIPTION:
The present study is a single-ascending dose (SAD) and multiple-ascending dose (MAD) evaluation of RLS-0071 in healthy volunteers. This study is designed to evaluate the safety and tolerability of RLS-0071 administered by the intravenous (IV) route to healthy subjects as single- and multiple-ascending doses. Importantly, a SAD/MAD study in healthy subjects is critical to generate robust pharmacokinetic (PK) data using intensified PK sample collection, not feasible in a patient study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years, inclusive, at the time of Screening.
2. A female study subject must meet one of the following criteria: If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study intervention, during the study, and for at least 30 days after the last dose of the study intervention.

   a. An acceptable method of contraception includes one of the following: i. Abstinence from heterosexual intercourse ii. Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch) iii. Intrauterine device (with or without hormones) -OR- b. Agrees to use a double barrier method (eg, condom and spermicide) during the study and for at least 30 days after the last dose of the study intervention Female subjects who are not of childbearing potential are exempt from contraceptive requirements. To be considered of nonchildbearing potential female subjects must meet the following requirements: Must be surgically sterile (documented hysterectomy, tubal ligation, or bilateral salpingo-oophorectomy at least 3 months prior to Day 1) or postmenopausal (defined as 12 months from the time of last spontaneous menses). If necessary, a follicle-stimulating hormone (FSH) level > 35 IU/L at Screening will be considered confirmatory in the absence of a clear postmenopausal history.
3. A male study subject who engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (eg, condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study intervention.
4. Medically healthy on the basis of medical history, physical examination, and clinical laboratory testing in the opinion of the Investigator or designee.
5. Nonsmokers and nonusers of nicotine-containing products, including e-cigarettes, for at least 6 continuous months before the first dose of study intervention and for the duration of the study, to be confirmed by cotinine testing at Screening.
6. Negative drug/alcohol testing at Screening and Check-in (Day -1).
7. Vital signs (after semirecumbent for at least 5 minutes) that are within the following ranges at Screening and Check-in (Day -1):

   1. Systolic blood pressure (BP), 90 to 140 mmHg, inclusive
   2. Diastolic BP, 50 to 90 mmHg, inclusive
   3. Heart rate (HR), > 45 to ≤ 100 bpm
8. Weight ≤ 90 kg and body mass index (BMI) ≥ 18 and ≤ 30 kg/m2 at Screening.
9. Normal renal function, defined as estimated creatinine clearance (CrCl) > 90 mL/min (calculated using the Modification of Diet in Renal Disease [MDRD] formula) at Screening; an Investigator can determine based on clinical judgment whether a lower clearance rate can be accepted based on the muscle composition of the subject.
10. Willing and able to provide voluntary, written informed consent to participate in the study.
11. Able to communicate well with the Investigator and/or study site personnel and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Use of any prescription or over-the-counter (OTC) medications, herbal products (eg, St John's Wort, milk thistle), or supplements/vitamins within 14 days before dosing with study intervention and for the duration of the study, with the exception of those approved by the Investigator and Sponsor (eg, oral contraceptives, hormone replacement therapy).
2. Receipt of any investigational agent or treatment within 30 days or 5 half-lives, whichever is longer, prior to Screening.
3. Receipt of any protein- or antibody-based therapeutic agents (eg, growth hormones or monoclonal antibodies) within 3 months before dosing with study intervention.

   Note: Influenza and COVID-19 vaccine will be allowed if all doses in the regimen have been administered more than 21 days before dosing with study intervention.
4. History of any major surgery within 6 months before dosing with study intervention.
5. History of hepatic disease, or current clinically significant liver function test results, defined as alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin and fractionated bilirubin, and alkaline phosphatase (AP) > 1.5 × upper limit of normal (ULN) at Screening.

   Note: Isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%.
6. History of any clinically relevant or chronic psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, hematological, or gastrointestinal abnormality (eg, inflammatory bowel disease).
7. History of severe allergic/anaphylactic reaction.
8. Diagnosis or positive Screening test for antinuclear antibodies (ANA), anti-double-stranded deoxyribonucleic acid (DNA) antibodies (anti-dsDNA), anti-ribonucleoprotein antibodies (anti-RNP), anti-Sjögren's syndrome type A antibodies (anti-Ro/SSA), anti-Sjögren's syndrome type B antibodies (anti-La/SSB), anti-Smith antibodies (anti-SM), and anti-phospholipid antibodies.
9. Subjects with a history of autoimmune disease, glomerulonephritis, or vasculitis.
10. Known history of allergy to any component of study intervention including polyethylene glycol (PEG).
11. History of any active infection within 14 days dosing with study intervention, if deemed clinically significant by the Investigator and Sponsor.
12. Any acute illness within 30 days before dosing with study intervention.
13. History of warfarin use or International Normalized Ratio (INR) ≥ 1.5.
14. Has a history (within 2 years before the first dose of study intervention) of moderate or severe use disorder for any substance other than caffeine (based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition [DSM-5] criteria).
15. Diagnosis of or positive Screening result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV)-1 or HIV-2.
16. Positive COVID-19 test or any prior COVID-19 diagnosis.
17. Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism, or excretion of RLS-0071.
18. Presence of clinically significant electrocardiogram (ECG) finding (confirmed upon repeat testing) that, in the opinion of the Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results, as follows:

    1. QTcF > 450 msec for males and > 470 msec for females or low, or flat T-waves making measurement of the interval unreliable at Screening or check-in (Day -1)
    2. Other ECG abnormalities considered clinically relevant in the judgment of the Investigator
19. Concurrent conditions that could interfere with safety and/or tolerability measurements, as determined by the Investigator or a designee.
20. Pregnant and/or lactating.
21. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to Screening.
22. Plasma donation within 7 days of Screening.
23. Inability to tolerate IV administration.
24. Poor venous access, as determined by the Investigator or a designee.
25. Unable or unwilling to cooperate with the site staff for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From initiation of study treatment (Day 1) through follow-up period (Day 30)
  Safety and tolerability will be assessed throughout the study by monitoring and evaluating TEAEs, including any complications resulting from the IV infusion. All AEs will be collected from the start of study intervention administration through Day 30 or Early Termination (ET). Adverse event grading will be defined by the CTCAE (latest version).
Incidence of abnormal laboratory test results | From initiation of study treatment (Day 1) through follow-up period (Day 30)

SECONDARY OUTCOMES:
Plasma maximum measured drug concentration (Cmax) | 0 - 1 week
Time of maximum concentration (Tmax) | 0 - 1 week
Area under the concentration-time curve (AUC) | 0 - 1 week
Terminal elimination half-life (T 1/2) | 0 - 1 week
Pharmacodynamic parameter - mCH50 assay | 0 - 1 week
  mCH50 assay for detection of inhibition of classical complement pathway activation
Pharmacodynamic parameter - C1q levels | 0 - 1 week

OTHER OUTCOMES:
Exploratory Biomarker - Membrane-attack complex assay (sC5b-9) | 0 - 1 week
Immunogenicity characteristics - presence of anti-RLS-0071 antibody (ADA) | From initiation of study treatment (Day 1) through follow-up period (Day 30)

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Cunnion, MD, Study Director — Chief Medical Officer, ReAlta Life Sciences, Inc.
Locations (1):
- Altasciences, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No